CLINICAL TRIAL: NCT01484821
Title: Assessment of in Vivo Skeletal Muscle Viscoelasticity (ARFI Imaging) With Aging and Cancer
Acronym: CAPARFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2011/29
Record Dates: First submitted 2011-11-22; First posted 2011-12-02 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; ARFI; DEXA; Cancer
MeSH Terms: conditions — Sarcopenia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Active Comparator): Volunteers (18 -30 years)
  Interventions: Device: ARFI
- Arm B (Active Comparator): Volunteers (70 years or older)
  Interventions: Device: ARFI
- Arm C (Experimental): 70 years patient or older with curative cares for cancer
  Interventions: Device: ARFI

INTERVENTIONS:
Device: ARFI — Muscle sonoelastography using ARFI(Acoustic Radiation Force Impulse) imaging

SUMMARY:
Sarcopenia is known to be associated with loss in muscle mass that results from a reduced number of muscle fibres, an atrophy of remaining muscle fibres, and an increased infiltration of non-contractile tissue (collagen, fat). Accentuated by cancer and treatments, sarcopenia impairs muscle function resulting in a higher risk of physical disability and death. The commonly used test for sarcopenia screening consists in a DEXA (Dual energy X-ray absorptiometry) scan. However, this test can't provide structural muscle information. In contrast, the mechanical properties of muscle tissue can be explored using an acoustic radiation force impulse (ARFI). The question remains whether muscle sonoelastography using ARFI imaging could be helpful for sarcopenia screening.

For this, volunteers will be recruited in three groups: ≤ 30 years (Gr A) and ≥ 70years, both without any serious chronic disease, and patients ≥ 70 years presenting curative cares for cancer (Gr C).

The volunteers belonging to the groups A and B will be followed during one day. The patients included in the group C will be followed during 6 months. For this latter group; the first visit (t0) will take place before treatment and the second visit will take place 6 months later (t6months) Volunteers will have clinical examinations (weight, stature, BMI, performance status/ ECOG) and will be evaluated on their nutritional status (MNA-SF, 24h dietary recall) and physical capacities (IPAQ, SPPB, lower limb muscle strength, 6-min walk test, QLQ-C30 items relative to the fatigue symptom).

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years old or more,
* Able to understand the protocol and to give their written consent,
* Health insurance.

Specific inclusion criteria:

* Group A: volunteers 18 to 30 yrs; without any pathology,
* Group B: volunteers ≥ 70 yrs; without any pathology,
* Group C: Performance status (ECOG) < 4; patients included in CAPADOGE study presenting curative cares for cancer by chemotherapy and/ or surgery and/or hormonotherapy and/or radiotherapy.

Exclusion Criteria:

* Intense activity in 7 preceding days,
* Functional dependency,
* under a legal protection.

Specific non-inclusion criteria:

* Groups A & B: serious chronic disease,
* Group C: Palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Viscoelasticity of the contracted Tibialis anterior muscle | Day 1 (group A, B and C) and month 6 (group C only)
  Describe and compare the distribution curves of viscoelasticity of the contracted Tibialis anterior muscle, measured by the ARFI shear wave velocity, between each group.

SECONDARY OUTCOMES:
Viscoelasticity of the contracted and relaxed Rectus femoris and Soleus muscles | Day 1 (group A, B and C) and month 6 (group C only)
Distribution curves of subcutaneous thickness in relaxed condition between each group on Rectus femoris and Soleus muscles | Day 1 (group A, B and C) and month 6 (group C only)
Compare fort each muscle the distribution curves of pennation angles in relaxed and contracted conditions between each group on Rectus femoris and Soleus muscles | Day 1 (group A, B and C) and month 6 (group C only)
Evaluate the influence of physical and/or nutritional status, age, and cancer pathology | Day 1 (group A, B and C) and month 6 (group C only)
Evaluate the intra-operator reproducibility | Day 1 (group A, B and C)

CONTACTS AND LOCATIONS:
Overall Officials: Nora FRULIO, Dr, Principal Investigator — University Hospital, Bordeaux, France
Locations (2):
- France (2):
  - CHU Bordeaux - Hôpital Saint André, Bordeaux
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac